CLINICAL TRIAL: NCT03025360
Title: Expanded Access to Provide Larotrectinib (LOXO-101) for the Treatment of Cancers With a NTRK Gene Fusion
Brief Title: Expanded Access to Provide Larotrectinib for the Treatment of Cancers With a NTRK Gene Fusion
Status: Approved for marketing | Type: Expanded Access
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20366
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Tumors Harboring NTRK Fusion
Keywords: Neurotrophic tyrosine receptor kinase (NTRK); NTRK1; NTRK2; NTRK3; Fusion Positive
MeSH Terms: interventions — larotrectinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Larotrectinib (Vitrakvi, BAY2757556) — Larotrectinib will be administered orally as capsule or liquid solution as specified by the treating physician.
  Other Names: LOXO-101

SUMMARY:
Larotrectinib expanded access is for patients with cancer with a NTRK1, NTRK2, or NTRK3 gene fusion, who are ineligible for an ongoing larotrectinib clinical trial or have other considerations that prevent access to larotrectinib through an existing clinical trial. Gene fusion occurs when a gene is made by joining parts of two different genes. NTRK gene fusion can lead to the development of solid tumors in a variety of tissue types. The study drug larotrectinib blocks the action of the NTRK gene fusion.

Expanded access is intended to treat individual patients with different types of cancers with a NTRK gene fusion who are unresponsive to current standard treatment for their condition and also are unable to participate in ongoing clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer with a NTRK1, NTRK2, or NTRK3 gene fusion
* Subjects are unable to participate in an ongoing larotrectinib clinical trial
* Medically suitable for treatment with larotrectinib

Exclusion Criteria:

* Currently enrolled in an ongoing clinical study of larotrectinib or another TRK inhibitor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult